CLINICAL TRIAL: NCT03424382
Title: CREATION Health Readmission Risk Assessment Tool
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1004998
Record Dates: First submitted 2018-01-23; First posted 2018-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure; COPD; Myocardial Infarction; Coronary Artery Bypass Graft; Pneumonia; Total Knee Replacement; Total Hip Replacement; Stroke
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Myocardial Infarction; Pneumonia; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase I: Participants will complete an intake form and assessment tool survey on an electronic device provided by research staff in their hospital room. If an individual is unable to complete the instrument, he or she may have another individual enter his or her answers on the electronic device.
- Phase II: Participants will complete an intake form and assessment tool survey on an electronic device provided by research staff in their hospital room. If an individual is unable to complete the instrument, he or she may have another individual enter his or her answers on the electronic device.

SUMMARY:
This study occurs in two phases. Phase 1 involves initial item development and measurement validation of a new tool for identifying hospitalized patients at high risk for preventable readmission. Primary tasks include item construction and content validation, data collection, analysis, and instrument refinement. Phase 2 involves administering the refined instrument to a new group of patients to determine final item content for the instrument, its factor structure, and its predictive validity.

DETAILED DESCRIPTION:
Participants will complete the instrument on an electronic device provided by research staff in the hospital room. If an individual is unable to complete the instrument, the participant may have another individual input answers on the electronic device. Hospitalized patients (n = 1240: 620 in Phase 1 and 620 in Phase 2) with a variety of chronic diseases will be recruited into the study. Study coordinators will recruit participants with the following diagnoses: heart failure, chronic obstructive pulmonary disease, acute myocardial infarction, coronary artery bypass graft, pneumonia, total knee or hip replacement, and stroke. These diagnoses were chosen because of the frequency with which patients are readmitted after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary admission diagnosis of heart failure, chronic obstructive pulmonary disease, acute myocardial infarction, coronary artery bypass graft, pneumonia, total knee or hip replacement, or stroke.
* Age 21 and over
* Able to provide informed consent
* Able to speak and read English
* Able to complete an electronic survey or relay answers to questions to another party who may complete the survey for the participant
* Resides in Central Florida and anticipates continued residence in Central Florida for the next 120 days
* Planned discharge to a non-hospital or residential care environment

Exclusion Criteria:

* Under age 21
* Does not speak or read English
* Permanent residence is outside Central Florida
* Not of cognitive capacity to provide valid responses
* Dementia or cognitive impairment that renders subject unable to provide informed consent
* Prescribed a known psychoactive medication that might reasonably affect the ability of the participant to provide valid responses

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients at Florida Hospital Orlando with one of the targeted diagnoses
Sampling Method: Probability Sample
Enrollment: 1218 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Social Determinant Survey Responses | 24 Months
  An Investigator developed measurement instrument (survey) will be used to gather participant self reported responses to questions regarding spirituality, nutrition, sleep, activity level, interpersonal relationships, home environment and access to transportation. Participants will be provided a five point Likert Scale to express agreement or disagreement with the questions.

SECONDARY OUTCOMES:
Readmission Status | 24 Months
  Data extraction from each participant's medical record will be used to determine the number of readmissions within 120 days post discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Robinson, Principal Investigator — Center for CREATION Health Research
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baltodano PA, Webb-Vargas Y, Soares KC, Hicks CW, Cooney CM, Cornell P, Burce KK, Pawlik TM, Eckhauser FE. A validated, risk assessment tool for predicting readmission after open ventral hernia repair. Hernia. 2016 Feb;20(1):119-29. doi: 10.1007/s10029-015-1413-2. Epub 2015 Aug 19. PMID 26286089
- [Background] Banoff KM, Milner K, Rimar J, Greer AE, Canavan M. Assessment of a Novel Tool for Identifying Hospitalized Patients with Heart Failure at Risk for 30-Day Readmission, High Cost, and Longer Length of Stay. Nurs Econ. 2016 Jul-Aug;34(4):172-81. PMID 29975022
- [Background] Floyd, F. J., & Widaman, K. F. (1995). Factor analysis in the development and refinement of clinical assessment instruments. Psychological Assessment, 7 (3), 286-299.
- [Background] Gorsuch, R. L. (1983). Factor analysis (2nd edition). New York: Laurence Earlbaum.
- [Background] Jencks SF, Williams MV, Coleman EA. Rehospitalizations among patients in the Medicare fee-for-service program. N Engl J Med. 2009 Apr 2;360(14):1418-28. doi: 10.1056/NEJMsa0803563. PMID 19339721
- [Background] Kansagara D, Englander H, Salanitro A, Kagen D, Theobald C, Freeman M, Kripalani S. Risk prediction models for hospital readmission: a systematic review. JAMA. 2011 Oct 19;306(15):1688-98. doi: 10.1001/jama.2011.1515. PMID 22009101
- [Background] National Medicare readmission findings: Recent data and trends. Centers for Medicare and Medicaid Services [Internet]. 2012. Available from: http://www.academyhealth.org/files/2012/sunday/ brennan.pdf.
- [Background] Naylor MD, Brooten DA, Campbell RL, Maislin G, McCauley KM, Schwartz JS. Transitional care of older adults hospitalized with heart failure: a randomized, controlled trial. J Am Geriatr Soc. 2004 May;52(5):675-84. doi: 10.1111/j.1532-5415.2004.52202.x. PMID 15086645
- [Background] Report to the congress: Promoting greater efficiency in Medicare. Medicare Payment Advisory Commission [Internet]. 2007 June 2007. Available from: http://www.caretransitions.org/documents/ MedPAC%20report.pdf.
- [Background] Rubin DJ, Handorf EA, Golden SH, Nelson DB, McDonnell ME, Zhao H. DEVELOPMENT AND VALIDATION OF A NOVEL TOOL TO PREDICT HOSPITAL READMISSION RISK AMONG PATIENTS WITH DIABETES. Endocr Pract. 2016 Oct;22(10):1204-1215. doi: 10.4158/E161391.OR. PMID 27732098
- [Background] Stauffer BD, Fullerton C, Fleming N, Ogola G, Herrin J, Stafford PM, Ballard DJ. Effectiveness and cost of a transitional care program for heart failure: a prospective study with concurrent controls. Arch Intern Med. 2011 Jul 25;171(14):1238-43. doi: 10.1001/archinternmed.2011.274. PMID 21788541
- [Background] Tabachnick, B. G., & Fidell, L. S. (2007). Using multivariate statistics (5th edition). Boston: Pearson Press.